CLINICAL TRIAL: NCT02382770
Title: International Register of Open Abdomen
Acronym: IROA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Principal Investigator, Federico Coccolini, MD, M.D., A.O. Ospedale Papa Giovanni XXIII
Other Study IDs: 15-15
Record Dates: First submitted 2015-02-27; First posted 2015-03-09 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Open Abdomen Procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (1):
- Open Abdomen patients: All patients underwent to open abdomen procedure
  Interventions: Procedure: Open abdomen procedure

INTERVENTIONS:
Procedure: Open abdomen procedure — Patients who may need at the end of surgical procedure will be left with open abdomen dressed with different devices or dressing according to the institutional indications.

SUMMARY:
To evaluate the different indications to Open Abdomen, the different techniques used to perform it, it's management, it's definitive closure and mortality rates linked to the different variables. Moreover to evaluate the 1 month and 1 year follow up in patients underwent to Open Abdomen.

ELIGIBILITY:
Inclusion Criteria:

* No age limit
* Indication to Open Abdomen
* Informed consent

Exclusion Criteria:

* Informed consent refusal
* No indication to Open Abdomen

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who may require to be undergone to open abdomen procedure
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Indications to open abdomen | Enrollment
Techniques to perform open abdomen | Enrollment
Management of open abdomen | Visit 2
Definitive closure techniques | Visit 4

SECONDARY OUTCOMES:
Mortality rates linked to different techniques of open abdomen | During All study period
Morbidity rates linked to different techniques of open abdomen | During All study period

CONTACTS AND LOCATIONS:
Overall Officials: Federico Coccolini, MD, Principal Investigator — Papa Giovanni XXIII, P.zza OMS 1, 24128 Bergamo, Italy
Locations (4):
- - Emergency and Trauma Surgery dept., Virginia Commonwealth University, Richmond, Virginia, United States
- Letterkenny Surgery dept. Letterkenny Hospital, Letterkenny, Ireland
- Italy (2):
  - Papa Giovanni XXIII hospital,, Bergamo
  - Emergency Surgery, Parma Universitary hospital, Parma

REFERENCES:
- [Derived] Sibilla MG, Cremonini C, Portinari M, Carcoforo P, Tartaglia D, Cicuttin E, Musetti S, Strambi S, Sartelli M, Radica MK, Catena F, Chiarugi M, Coccolini F; IROA Study Group. Patients with an Open Abdomen in Asian, American and European Continents: A Comparative Analysis from the International Register of Open Abdomen (IROA). World J Surg. 2023 Jan;47(1):142-151. doi: 10.1007/s00268-022-06733-4. Epub 2022 Nov 3. PMID 36326921
- [Derived] Coccolini F, Gubbiotti F, Ceresoli M, Tartaglia D, Fugazzola P, Ansaloni L, Sartelli M, Kluger Y, Kirkpatrick A, Amico F, Catena F, Chiarugi M; IROA study group. Open Abdomen and Fluid Instillation in the Septic Abdomen: Results from the IROA Study. World J Surg. 2020 Dec;44(12):4032-4040. doi: 10.1007/s00268-020-05728-3. Epub 2020 Aug 24. PMID 32833107
- [Derived] Ceresoli M, Salvetti F, Kluger Y, Braga M, Vigano J, Fugazzola P, Sartelli M, Ansaloni L, Catena F, Coccolini F; IROA study group. Open Abdomen in Obese Patients: Pay Attention! New Evidences from IROA, the International Register of Open Abdomen. World J Surg. 2020 Jan;44(1):53-62. doi: 10.1007/s00268-019-05209-2. PMID 31602518
- [Derived] Coccolini F, Montori G, Ceresoli M, Catena F, Ivatury R, Sugrue M, Sartelli M, Fugazzola P, Corbella D, Salvetti F, Negoi I, Zese M, Occhionorelli S, Maccatrozzo S, Shlyapnikov S, Galatioto C, Chiarugi M, Demetrashvili Z, Dondossola D, Yovtchev Y, Ioannidis O, Novelli G, Nacoti M, Khor D, Inaba K, Demetriades D, Kaussen T, Jusoh AC, Ghannam W, Sakakushev B, Guetta O, Dogjani A, Costa S, Singh S, Damaskos D, Isik A, Yuan KC, Trotta F, Rausei S, Martinez-Perez A, Bellanova G, Fonseca VC, Hernandez F, Marinis A, Fernandes W, Quiodettis M, Bala M, Vereczkei A, Curado RL, Fraga GP, Pereira BM, Gachabayov M, Chagerben GP, Arellano ML, Ozyazici S, Costa G, Tezcaner T, Ansaloni L. IROA: International Register of Open Abdomen, preliminary results. World J Emerg Surg. 2017 Feb 21;12:10. doi: 10.1186/s13017-017-0123-8. eCollection 2017. PMID 28239409
- [Derived] Coccolini F, Catena F, Montori G, Ceresoli M, Manfredi R, Nita GE, Moore EE, Biffl W, Ivatury R, Whelan J, Fraga G, Leppaniemi A, Sartelli M, Di Saverio S, Ansaloni L. IROA: the International Register of Open Abdomen.: An international effort to better understand the open abdomen: call for participants. World J Emerg Surg. 2015 Aug 16;10:37. doi: 10.1186/s13017-015-0029-2. eCollection 2015. PMID 26279673